CLINICAL TRIAL: NCT02042638
Title: The Effects of Gonadotropin Replacement Therapy in Patients With Hypogonadism
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Aydogan Aydogdu, MD, Gulhane School of Medicine
Other Study IDs: 27122013
Record Dates: First submitted 2013-12-28; First posted 2014-01-23 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2013-12

CONDITIONS: Idiopathic Hypogonadotropic Hypogonadism
MeSH Terms: conditions — Idiopathic Hypogonadotropic Hypogonadism | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 16 treatment naive Hypogonadotropic hypogonadism patients: Treatment naive 16 patients with idiopathic hypogonadotrophic hypogonadism
  Interventions: Drug: hCG 1500 IU three times a week; Drug: Pregnyl (hCG) ampule 1500 IU/three times a week

INTERVENTIONS:
Drug: hCG 1500 IU three times a week
  Other Names: Pregnyl (Organon) ampule 1500 IU
Drug: Pregnyl (hCG) ampule 1500 IU/three times a week

SUMMARY:
Effects of hCG replacement therapy on metabolic syndrome parameters in hypogonadotrophic hypogonadism.

ELIGIBILITY:
Inclusion Criteria: Serum testosterone concentration < 300ng/dL Absence of a pituitary or hypothalamic mass lesions, Presence of gonadotropin response to GnRH, -

Exclusion Criteria: Previous androgen treatment, diabetes mellitus, arterial hypertension other hormone deficiencies

-

Ages: 16 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Idiopathic Hypogonadotropic Hypogonadism
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
HDL after hCG treatment | 2011-2013
  2011-2013
LDL levels after hCG treatment | 2011-2013
total cholesterole levels after hCG treatment | 2011-2013

SECONDARY OUTCOMES:
Body fat ratio after hCG treatment | 2011-2013
hsCRP levels after hCG treatment | 2011-2013

CONTACTS AND LOCATIONS:
Overall Officials: Fahri Bayram, Proffesor, Study Director — Erciyes University School of Medicine Depatment of Endocrinology and Metabolism Kayseri TURKEY
Locations (1):
- Gulhane School of Medicine Dep. of Endocrinology and Metabolism, Ankara, Turkey (Türkiye)